CLINICAL TRIAL: NCT02320812
Title: A Prospective, Multicenter, Open-Label, Single-Arm Study of the Safety and Tolerability of a Single, Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects With Retinitis Pigmentosa (RP)
Brief Title: Safety of a Single, Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: jCyte, Inc (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JC-01
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Retinitis Pigmentosa (RP)
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated subjects (Experimental): human retinal progenitor cells
  Interventions: Biological: human retinal progenitor cells

INTERVENTIONS:
Biological: human retinal progenitor cells — single intravitreal injection of 0.5 - 3.0 million human retinal progenitor cells (hRPC)
  Other Names: jCell

SUMMARY:
This study evaluates the safety and potential activity of a single dose of live human retinal progenitor cells (jCell) administered to adults with retinitis pigmentosa. Four different dose levels of cells will be assessed in each of two groups of patients.

DETAILED DESCRIPTION:
The primary purpose of this study is to test the safety and tolerability of the administration of a single dose of jCell to adults with retinitis pigmentosa.

The goal of jCell therapy is to preserve vision by intervening in the disease at a time when host photoreceptors can be protected and potentially reactivated.

Human allogeneic retinal progenitor cells will be injected into adults with advanced RP to see if the procedure is safe, if the cells survive, and whether they have any impact on the visual status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RP confirmed by electroretinogram (ERG) and willing to consent to mutation typing, if not already done
* Best corrected visual acuity (BCVA) 20/63 or worse and no worse than hand motions (HM)
* Adequate organ function and negative infectious disease screen
* Female of childbearing potential must have negative pregnancy test and be willing to use medically accepted methods of contraception throughout the study

Exclusion Criteria:

* Eye disease other than RP that impairs visual function
* Pseudo-RP, cancer-associated retinopathies
* History of malignancy or other end-stage organ disease, or any chronic disease requiring continuous treatment with system steroids, anticoagulants or immunosuppressive agents
* Known allergy to penicillin or streptomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Kuppermann, MD, Principal Investigator — Gavin Herbert Eye Institute, UCI, Irvine, CA
Locations (2):
- United States (2):
  - The Gavin Herbert Eye Institute, Univ California Irvine, Irvine, California
  - Retina-Vitreous Associates Medical Group, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang J, Kuppermann BD, Liao D, Mehta MC, Hsiang C, Menges S, Boyer DS, Klassen H. Retinal progenitor cells (jCell) for retinitis pigmentosa. Front Cell Neurosci. 2025 Aug 25;19:1646156. doi: 10.3389/fncel.2025.1646156. eCollection 2025. PMID 40927136

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treated Subjects
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treated Subjects
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability
Description: proportion of subjects with treatment emergent adverse events (TEAE), related TEAE and severe TEAE
Time Frame: 12 months
Population: all treated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Subjects
Number analyzed (Participants) | 28
Participants
  Subjects with TEAE | 25
  Subjects with related TEAE | 21
  Subjects with grade 3 TEAE | 1

2. Secondary Outcome: Change in Mean Best Corrected Visual Acuity (BCVA)
Description: change in mean best corrected visual acuity in test eye versus untreated eye; BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. Change between baseline and month 12 is reported.
Time Frame: 12 months
Population: all treated subjects
Measure: Mean (Full Range); unit: number of letters read correctly
Groups:
- 0.5 Million Cells Cohort: subjects who received 0.5 million human retinal progenitor cells (hRPC)
- 1.0 Million Cells Cohort: subjects who received 1.0 million hRPC
- 2.0 Million Cells Cohort: subjects who received 2.0 million hRPC
- 3.0 Million Cells Cohort: subjects who received 3.0 million hRPC
Arm/Group | 0.5 Million Cells Cohort | 1.0 Million Cells Cohort | 2.0 Million Cells Cohort | 3.0 Million Cells Cohort
Number analyzed (Participants) | 8 | 8 | 6 | 6
number of letters read correctly | 1.4 [-3 to 11] | 1.0 [-3 to 11] | 4.8 [0 to 8] | 9.0 [0 to 12]

ADVERSE EVENTS:
Time Frame: one year following single intravitreal injection of hRPC
Arm/Group | Treated Subjects
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=28)
migratory pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=28)
anterior chamber flare (Eye disorders) | 5 (5)
conjunctival hemorrhage (Eye disorders) | 10 (10)
eye pain (Eye disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT02320812/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT02320812/SAP_001.pdf